CLINICAL TRIAL: NCT05678777
Title: Use of Galvanic Skin Response(GSR) to Measure Peripheral Block Activity
Brief Title: Use of Galvanic Skin Response to Measure Peripheral Block Activity
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Adiyaman University (Other)
Responsible Party: Principal Investigator, Fikret Ozerdem, assistant doctor, Adiyaman University
Other Study IDs: 18/01/2022-2022/1-10; Fadime Tosun (Other: Adiyaman University)
Record Dates: First submitted 2023-01-02; First posted 2023-01-10 (Actual); Last update posted 2023-01-10 (Actual); Status verified 2023-01

CONDITIONS: Regional Anesthesia
Keywords: Galvanic Skin Response; Peripheral Block
MeSH Terms: interventions — Galvanic Skin Response

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Galvanic Skin Response — The probe will be attached to the patient's finger and the Galvanic Skin Response will be measured

SUMMARY:
the investigators aim in this study is to determine whether the block is successful in successful infraclavicular brachial plexus blocks performed with USG, according to the change in GSR value in the upper extremity blocked due to sympathetic nerve blockade. Block success will be evaluated by sensory and motor examination of the blocked arm.

DETAILED DESCRIPTION:
Peripheral nerve block is one of the commonly used blocks in regional anesthesia. In regional anesthesia applications, there are important advantages such as being conscious of the patient, expressing his complaints, continuation of spontaneous breathing, preservation of airway reflexes, continuation of analgesia in the postoperative period and early mobilization of the patient.

In 1978, ultrasound (USG) was used for the first time in peripheral nerve block. With USG, it is possible to monitor the nerves and anatomical structures, follow the needle, and reduce the dose by monitoring the distribution of the local anesthetic administered. Therefore, USG-guided peripheral nerve blocks are frequently used in anesthesia practice.

The Galvanic Skin Response (GSR) is a simple way to obtain autonomic nervous system dependent sweat gland function as a parameter.

Physically, the galvanic skin response is the change in the electrical structure of the skin to various stimuli. Changes in tension measured from the skin surface are recorded. The galvanic skin response is a useful, simple and reproducible electrophysiological technique for investigating sympathetic nervous system function.

The relaxation, calming response that accompanies an increase in skin resistance (causing a decrease in GSR meter) is the body's combat response that accompanies a decrease in skin resistance (causing an increase in GSR meter). Generally, low conductivity is a sign of relaxation. High conductivity is a sign of emotional, mental, or physical arousal. The galvanic skin response is a simple way to obtain autonomic nervous system-related sweat gland function as a parameter.

the investigators aim in this study is to determine whether the block is successful in successful infraclavicular brachial plexus blocks performed with USG, according to the change in GSR value in the upper extremity blocked due to sympathetic nerve blockade. Block success will be evaluated by sensory and motor examination of the blocked arm. The relaxation, calming response that accompanies an increase in skin resistance (causing a decrease in GSR meter) is the body's combat response that accompanies a decrease in skin resistance (causing an increase in GSR meter). Generally, low conductivity is a sign of relaxation. High conductivity is a sign of emotional, mental, or physical arousal.

In the investigators clinic, peripheral nerve blocks accompanied by USG are frequently used in anesthesia practice.

OBJECTİVE: Successful peripheral nerve blockade results in local vasodilation, increased local blood flow, and some increase in skin temperature due to sympathetic fiber blocking. However, in busy operating room conditions, these clinical signs may not appear quickly enough to confirm block adequacy, especially before or during surgery, and may not be used for clinical decision making. Traditional methods for assessing block success are time consuming and require patient cooperation. For the success of the block, it is aimed to use the Galvanic Skin Response (GSR) value, which is a non-invasive method that does not require patient cooperation and provides rapid evaluation.

Galvanic Skin Response (GSR) measurement is a non-invasive and rapid assessment that allows us to observe the skin resistance change with two probes attached to the fingertip. In the investigators study, we aimed to show that the Galvanic Skin Response (GSR) measurement method is a reliable and objective method to evaluate the adequacy of peripheral nerve blocks.

METHODS: This research; It is a prospective observational study. In patients who have performed infraclavicular brachial plexus block; The correlation of Galvanic skin response (GSR) values measured with the finger probe that we attached to the patient's two fingers before and after the block, with the success of the block will be examined. the investigators study is not invasive, it is only in the form of examining finger probe measurements and will not create an additional cost for the investigators hospital and the participants..

ELIGIBILITY:
Inclusion Criteria:

1. ASA1-ASA2 patients
2. Patients between the ages of 18-65
3. Patients who underwent infraclavicular block

Exclusion Criteria:

1. ASA3-ASA4 patients
2. Patients younger than 18 years old and over 65 years old
3. Patients who do not want to be included in the study
4. Patients in whom infraclavicular brachial plexus block is contraindicated
5. Patients who cannot cooperate
6. Those with diabetes mellitus
7. Patients who have failed infraclavicular brachial plexus block and switched to general anesthesia
8. Those with peripheral artery disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients aged 18-65 who will undergo upper extremity surgery
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-01-30 (Actual); Primary Completion 2023-02-28 (Estimated); Study Completion 2023-03-30 (Estimated)

PRIMARY OUTCOMES:
Galvanic Skin Response | 30/01/2023-28/02/2023

CONTACTS AND LOCATIONS:
Locations (1):
- Adiyaman University, Adıyaman, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
ı am undecided about sharing individual participant data with other researchers

REFERENCES:
- [Background] Tarvainen MP, Koistinen AS, Valkonen-Korhonen M, Partanen J, Karjalainen PA. Analysis of galvanic skin responses with principal components and clustering techniques. IEEE Trans Biomed Eng. 2001 Oct;48(10):1071-9. doi: 10.1109/10.951509. PMID 11585030
- [Result] Marhofer P, Greher M, Kapral S. Ultrasound guidance in regional anaesthesia. Br J Anaesth. 2005 Jan;94(1):7-17. doi: 10.1093/bja/aei002. Epub 2004 Jul 26. PMID 15277302